CLINICAL TRIAL: NCT02579707
Title: A Phase 1, Open-Label, Randomized, 2-Period Crossover Study To Evaluate The Effect Of Food On AG-120 Pharmacokinetics Following Single Oral Dose Administration To Healthy Subjects
Brief Title: Food Effect Study of AG120 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AG120-C-004
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: Unfed (Active Comparator): Treatment A: Single oral dose of AG-120 at Hour 0 on Day 1, following a 10-hour overnight fast.
  Interventions: Drug: AG120
- Treatment B: Fed (Active Comparator): Treatment B: Single oral dose of AG-120 at Hour 0 on Day 1, 30 minutes after the start of a high-fat breakfast.
  Interventions: Drug: AG120
- Part 2 Single Dose (Experimental): PART 2 is an open-label study to determine the safety and PK parameters of a single 1000-mg oral dose of AG-120.
  Interventions: Drug: AG120

INTERVENTIONS:
Drug: AG120 — AG120 in fed and fasted conditions. Part 2- AG120 single dose exposure

SUMMARY:
This will be a 2-part study. PART 1 is an open-label, randomized, food effect study of AG-120. Subjects will be enrolled to a fed/fasted or fasted/fed treatment sequence in a 2-period crossover design. PART 2 is an open-label study to determine the safety and PK parameters of a single 1000-mg oral dose of AG-120.

ELIGIBILITY:
Inclusion Criteria:

1. males or females, aged 18 to 55 years, inclusive
2. within body mass index (BMI) range of 18 to 33 kg/m2, inclusive
3. in good health, determined by absence of clinically significant findings from medical history, 12-lead ECG, and vital signs
4. fasted clinical laboratory values within the normal reference range for the test laboratory, unless deemed not clinically significant by the Investigator. (Calcium, magnesium, and potassium levels within normal ranges)
5. negative test for selected drugs of abuse and cotinine at Screening (does not include alcohol) and at Check-in of Period 1 (Parts 1 and 2) and Period 2 (Part 1) (does include alcohol via breathalyzer)
6. negative hepatitis panel (including hepatitis B surface antigen and hepatitis C virus antibody) and negative human immunodeficiency virus (HIV) antibody screens
7. female subjects with reproductive potential must agree to undergo medically supervised pregnancy test prior to study drug administration. Pregnancy tests will be performed at Screening and confirmed negative at each Check-in
8. females of reproductive potential must agree to abstain from sexual intercourse or to use 2 highly effective forms of contraception from the time of giving informed consent, during the study, and for 90 days following the last dose of AG-120.
9. males must either be sterile or agree to use 2 of the following approved methods of contraception from time of giving informed consent until 90 days following the last dose administration. Subjects will refrain from sperm donation from time of giving informed consent until 90 days following the last dose administration
10. able to comprehend and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

1. history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator)
2. history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator
3. history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy and hernia repair will be allowed
4. history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant. QTcF values must be within ranges indicated in inclusion criteria #3
5. history of alcoholism or drug addiction within 2 years before first dose administration, or positive drug screening test reflecting consumption of illicit drugs or positive alcohol screen at each Check-in
6. use of any tobacco- or nicotine-containing products (including but not limited to cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to Screening through Study Completion, or positive cotinine screen at Screening or each Check-in
7. unwilling to refrain from strenuous exercise from 48 hours prior to each Check-in and during the period of confinement at the Clinical Research Unit and otherwise maintain their normal level of physical activity throughout the entire study (ie, will not begin a new exercise program nor participate in any unusually strenuous physical exertion)
8. participation in any other clinical trial in which an investigational study drug was administered within 5 half-lives or 30 days from Screening, whichever is longer
9. use of hormonal oral, implantable, injectable, or transdermal contraceptives from the time of signing the ICF (females only) until 90 days after the last dose administration
10. use of any prescription medications/products within 14 days prior to initial Check-in through Study Completion, unless deemed acceptable by the Investigator
11. use of any over-the-counter, nonprescription preparations including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations, within 7 days prior to initial Check-in through Study Completion, unless deemed acceptable by the Investigator
12. poor peripheral venous access
13. donation of blood or plasma within 8 weeks before first dose administration through Study Completion
14. receipt of blood products within 2 months prior to initial Check-in and for at least 28 days following the last dose of study drug
15. any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cmax | Day 1 predose (for each period as applicable) (0 hour [approximately 45 minutes prior to dose]) and 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 48, 72, 120, 168, 240, 336, and 504 hours post dose.
  Maximum observed concentration of AG-120
Incidence of adverse events | 22 days
  Assessment of adverse events
Tmax | Day 1 predose (for each period as applicable) (0 hour [approximately 45 minutes prior to dose]) and 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 48, 72, 120, 168, 240, 336, and 504 hours post dose.
  Time of maximum concentration of AG-120
AUC0-t | Day 1 predose (for each period as applicable) (0 hour [approximately 45 minutes prior to dose]) and 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 48, 72, 120, 168, 240, 336, and 504 hours post dose.
  Area under the concentration-time curve from Hour 0 to the last measurable concentration
AUC0-infinity | Day 1 predose (for each period as applicable) (0 hour [approximately 45 minutes prior to dose]) and 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 48, 72, 120, 168, 240, 336, and 504 hours post dose.
  Area under the concentration-time curve extrapolated to infinity
t1/2 | Day 1 predose (for each period as applicable) (0 hour [approximately 45 minutes prior to dose]) and 0.5, 1, 2, 3, 4, 6, 9, 12, 24, 48, 72, 120, 168, 240, 336, and 504 hours post dose.
  Apparent terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Sam Agresta, MD, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- Research Site, Madison, Wisconsin, United States